CLINICAL TRIAL: NCT05156853
Title: Sustainable Diets in Families in Copenhagen - Menus With Alternative Proteins Meals
Brief Title: Sustainable Diets in Families in Copenhagen
Acronym: SUSINCHAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Nanna Roos, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D229
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Insect Proteins
Keywords: Insect proteins; Alternative proteins; Human intervention study; Novel food acceptance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the taste and nature of the intervention foods, blinding of study staff and participants is not possible during this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insect-based menu (Experimental): Replacement of meat proteins with insect-based alternatives at main meals 3 times weekly.
  Interventions: Dietary Supplement: Insect menus
- Plant-based menu (Active Comparator): Replacement of meat proteins with plant-based alternatives at main meals 3 times weekly.
  Interventions: Dietary Supplement: Plant menus

INTERVENTIONS:
Dietary Supplement: Insect menus — The insect menus will consist of 6 different products: flatbread, spice-mix, paste, minced meat, sausage and falafels. The products are based on either crickets, mealworms or buffaloworm larvae.
  Arms: Insect-based menu
Dietary Supplement: Plant menus — The plant menus will be based on products which can be purchased in normal supermarkets and chosen to be as equal to the insect-based products as possible.
  Arms: Plant-based menu

SUMMARY:
SUSINCHAIN investigates the impact of exposing families (an adult and a child) to meals with alternative proteins (insect-based or plant-based products) on dietary pattern, intake of meat and total protein.

DETAILED DESCRIPTION:
The overall objective of this study is to investigate the impact of exposing paired participants (an adult and a child) to dinner menus of meals with alternative proteins (insect-based or plant-based products) on dietary pattern, intake of meat, and protein over a six-week intervention period. The insect-based menu is the experimental exposure and the plant-based menu is the positive control menu.

The hypothesis is that test menus of meals with alternative proteins will replace the meat consumed during dinner, resulting in maintaining the total protein intake while replacing 20% of the meat protein with alternative protein on a weekly basis.

The assumption is that the insect-based menus will replace meat protein similarly or to a larger extend than the positive control group receiving the comparable plant-based menu. The inclusion of the positive control group allows us to isolate the specific impact of exposure to insect-based menu from the exposure to dietary change of more familiar plant-based products.

The study is a randomized intervention trial recruiting 80 paired participants of an adult and a child age 8-10 year living together in a family, alone or with other family members. The paired participants are randomized to receive one of two menus of meals with alternative proteins, either plant-based or insect-based. Measurements (dietary records, questionnaires) as well as biological samples (urine collection) are taken primarily at baseline (week 0) and endline (week 6).

ELIGIBILITY:
This study recruits families in which one adult and one child are enrolled as participants.

Adults must:

* Be healthy.
* Determined from the self-reported medical history or when a clinical condition exists, when this is considered to be irrelevant (i.e. not influencing the safety for the participant or study outcomes) for the study by the study medical doctor.
* Eat meat for dinner at least 5 days a week in average.
* Be willing to consume insect- and plant-based foods.
* Be able to talk, read and understand Danish in order to understand the study procedures properly.
* Have basic computer competence.
* Have freezer capacity for two weeks of food.
* If the custody holders of a child, who wants to participant, do not want to participate, another adult from the household can participate. It is still the custody holders who are responsible for the child's participation in the study.

Children must:

* Be healthy.
* Determined from the self-reported medical history or when a clinical condition exists, when this is considered to be irrelevant (i.e. not influencing the safety for the participant or study outcomes) for the study by the study medical doctor.
* Eat meat for dinner at least 5 days a week in average.
* Age: 8-10 years.
* Be able to talk and understand Danish in order to understand the study procedures properly.
* Be willing to consume insect- and plant-based foods.

Exclusion Criteria (adult and child):

Individuals will be excluded if they have:

* Possess any food allergies or intolerances.
* Possess a dust mite allergy or intolerance.
* Follow one or more restricted diets (veganism, gluten-free, keto, vegetarianism, etc.).
* Use protein supplements, such as whey protein powder.
* Participation in other clinical studies.
* Gastrointestinal, kidney or liver disorders.
* Chronic inflammation disorders (excluding obesity).
* Diagnosed psychiatric disorder including depression requiring treatment, but can be accepted in judgement with the daily study manager, site-PI, PI or clinical responsible.
* Systematic antibiotic use < 1 month prior to the study.
* Lack of abilities (physical and psychological) to be complied with the procedures in the protocol, as evaluated by the daily study manager, site-PI, PI or clinical responsible.

Exclusion criteria related to adults:

* Pregnant or lactating within the study period.
* Self-reported use of drugs of abuse within the previous 12 months, including cannabis.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in intake of total daily amount of meat protein at baseline and endline | 6 weeks
  Data from 4 days dietary registration at each time-point
Change in proportion of meat protein of the total protein intake | 6 weeks
  Meat intake assessed by 4 day dietary registration, total protein intake assessed by 4 day dietary registration with biochemical validation by spot urine N excretion
Counts of main meals with meat and alternative protein products | 6 weeks
  Assessed during baseline week and each intervention week, including week of endline assessment

SECONDARY OUTCOMES:
Change in the sensory evaluation of the intervention foods | 6 weeks
  Changes in the sensory parameters for liking of the intervention food measured on Likert scale from 1 (extremely bad) to 7 (extremely good), meaning the higher score, the higher liking of the intervention food. Each paired participants are randomized to assess two of the six products at the first intervention week and the last intervention week.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen - Department of Nutrition, Exercise and Sports, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maya C, Wilderspin DE, Costa AIA, Cunha LM, Roos N. Introducing menus of three weekly insect- or plant-based dinner meals slightly reduced meat consumption in Danish families: Results of a randomized intervention study. Appetite. 2024 Dec 1;203:107689. doi: 10.1016/j.appet.2024.107689. Epub 2024 Oct 1. PMID 39357104
- [Derived] Maya C, Cunha LM, de Almeida Costa AI, Veldkamp T, Roos N. Introducing insect- or plant-based dinner meals to families in Denmark: study protocol for a randomized intervention trial. Trials. 2022 Dec 20;23(1):1028. doi: 10.1186/s13063-022-07000-6. PMID 36539897